CLINICAL TRIAL: NCT02981602
Title: A Phase 2, Double-Blinded, Randomized, Placebo-Controlled, Dose-Escalation Study to Examine the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of ISIS 505358 in Treatment-Naïve Patients With Chronic HBV Infection
Brief Title: Safety, Tolerability, Pharmacokinetics and Antiviral Activity of IONIS-HBVRx in Treatment-Naïve Patients With Chronic HBV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 205695; ISIS 505358-CS3 (Other: Ionis Pharmaceuticals, Inc.)
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Results first posted 2020-12-21 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis B; Chronic Hepatitis B Atypical
Keywords: Hepatitis; Chronic; HBV
MeSH Terms: conditions — Hepatitis B; Hepatitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IONIS-HBVRx (Experimental): Ascending multiple doses of IONIS-HBVRx by subcutaneous (SC) injection
  Interventions: Drug: IONIS-HBVRx
- Placebo (Placebo Comparator): Sterile Normal Saline (0.9% NaCl) calculated volume to match active comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IONIS-HBVRx — Ascending multiple doses of IONIS-HBVRx by subcutaneous (SC) injection
  Other Names: ISIS 505358
  Arms: IONIS-HBVRx
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To examine the safety and tolerability of IONIS-HBVRx administration to treatment-naive patients with chronic hepatitis B virus infection

DETAILED DESCRIPTION:
This study examines the effects of IONIS-HBVRx or placebo (3:1 randomization) administered subcutaneously to treatment-naïve patients who are chronically infected with HBV and the effects of subsequent nucleos(t)ide analogue treatment on these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Chronic HBV infection ≥6 months (e.g., positive for serum HBsAg ≥ 6 months)
* Plasma HBV DNA ≥ 2 x 1000 IU/mL (HBV DNA adequately suppressed for exploratory nucleos(t)ide analogue experienced cohort)
* Serum HBsAg ≥ 50 IU/mL
* Exploratory nucleos(t)ide analogue experienced cohort only: currently taking and have been taking tenofovir or entecavir without changes in drug, dose level and/or frequency of administration for ≥ 12 months and expect to continue taking without change through to the end of their participation in this study

Exclusion Criteria:

* Current or prior receipt of anti-HBV nucleos(t)ide analogue therapy. Patients who have failed prior interferon treatment, greater than 6 months prior to Screening, may be evaluated for possible participation in the study (not applicable for exploratory nucleos(t)ide analogue experienced cohort)
* History of liver cirrhosis and/or evidence of cirrhosis as determined by any of the following:

  1. Liver biopsy (i.e., Metavir Score F4) within 2 years of Screening, or
  2. Fibroscan > 12 KPa, within 12 months of Screening, or
  3. AST-to-Platelet Index (APRI) > 2 and Fibrosure result > 0.7 within 12 months of Screening For patients without a test for cirrhosis in the above timeframes, Fibroscan, or APRI and Fibrosure, may be performed during the screening period to rule out cirrhosis
* History of liver failure as evidenced by ascites, hepatic encephalopathy, and/or gastric or esophageal varices
* History of liver disease other than Hepatitis B
* Co-infection with hepatitis C virus (HCV), human immunodeficiency virus (HIV), or hepatitis D virus (HDV)
* BMI > 35 kg/m2
* History of, or suspected presence of vasculitis
* Received solid organ or bone marrow transplant
* Currently taking, or took within 3 months of Screening, any immunosuppressing drugs (e.g., prednisone)
* Diagnosed hepatocellular carcinoma or suspected hepatocellular carcinoma as evidenced by screening alpha-fetoprotein ≥ 200 ng/mL. If the screening alpha-fetoprotein is ≥ 50 ng/mL and < 200 ng/mL, the absence of liver mass must be documented by imaging within 6 months before randomization
* Clinically-significant abnormalities aside from chronic HBV infection in medical history (e.g., previous acute coronary syndrome within 6 months of Screening, major surgery within 3 months of Screening, uncontrolled diabetes) or physical examination
* History of bleeding diathesis or coagulopathy
* History of extrahepatic disorders possibly related to HBV immune complexes (e.g., glomerulonephritis, polyarteritis nodosa)
* History of excess alcohol consumption within 6 months of Screening
* History of drug abuse or dependence, or recreational use of drugs: within 3 months of Screening for soft drugs (such as marijuana) and within 1-year of Screening for hard drugs (such as cocaine, phencyclidine [PCP])

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Queen Mary Hospital, Hong Kong, Hong Kong
- South Korea (6):
  - Korea University Ansan Hospital, Ansan
  - Inje University Busan Paik Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Pusan National University Hospital, Pusan
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul

REFERENCES:
- [Derived] Yuen MF, Heo J, Jang JW, Yoon JH, Kweon YO, Park SJ, Tami Y, You S, Yates P, Tao Y, Cremer J, Campbell F, Elston R, Theodore D, Paff M, Bennett CF, Kwoh TJ. Safety, tolerability and antiviral activity of the antisense oligonucleotide bepirovirsen in patients with chronic hepatitis B: a phase 2 randomized controlled trial. Nat Med. 2021 Oct;27(10):1725-1734. doi: 10.1038/s41591-021-01513-4. Epub 2021 Oct 12. PMID 34642494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated safety, tolerability, pharmacokinetics and antiviral activity of GSK3228836 in two population of participants with Chronic Hepatitis B (CHB) virus infection: treatment-naive participants (Cohorts 1, 2 and 3) and participants on stable nucleos(t)ide treatment (Cohort 4)
Pre-assignment Details: A total of 31 participants were enrolled and received either GSK3228836 or placebo. In Cohort 3 participants were administered GSK3228836 300 milligram [mg] instead of 450 mg as per sponsor's decision, hence Cohort 2 and Cohort 3 have been combined.
Groups:
- Cohort 1 GSK3228836 150 mg: Treatment-naive participants were subcutaneously administered GSK3228836 150 mg on Days 1, 4, 8, 11, 15 and 22 by trained study center personnel in abdomen, upper arm or thigh.
- Cohort 2 and Cohort 3 GSK3228836 300 mg: Treatment-naive participants were subcutaneously administered GSK3228836 300 mg on Days 1, 4, 8, 11, 15 and 22 by trained study center personnel in abdomen, upper arm or thigh.
- Cohorts 1-3 Placebo: Treatment-naive participants were subcutaneously administered placebo on Days 1, 4, 8, 11, 15, and 22 by trained study center personnel in abdomen, upper arm or thigh.
- Cohort 4 GSK3228836 300 mg: Participants on stable nucleos(t)ide treatment were subcutaneously administered GSK3228836 300 mg on Days 1, 4, 8, 11, 15 and 22 by trained study center personnel in abdomen, upper arm or thigh.
- Cohort 4 Placebo: Participants on stable nucleos(t)ide treatment were subcutaneously administered placebo on Days 1, 4, 8, 11, 15 and 22 by trained study center personnel in abdomen, upper arm or thigh.
Period: Overall Study
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Started | 6 | 12 | 6 | 5 | 2
Completed | 6 | 12 | 6 | 4 | 2
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: In Cohort 3 participants were administered GSK3228836 300 mg instead of 450 mg as per sponsor's decision, hence Cohort 2 and Cohort 3 have been combined.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo | Total
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (11.22) | 42.6 (14.12) | 49.3 (12.66) | 48.4 (7.40) | 37.0 (2.83) | 44.5 (11.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 2 | 1 | 1 | 15
  Male | 3 | 4 | 4 | 4 | 1 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 6 | 12 | 6 | 5 | 2 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Non-Serious Adverse Events (Non-SAEs >=5%)
Description: An adverse event is any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product. Any adverse event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any important medical event according to medical judgment were categorized as SAE.
Time Frame: Up to Day 211
Population: Safety Population includes all randomized participants who received at least 1 dose of GSK3228836 or placebo. In Cohort 3 participants were administered GSK3228836 300 mg instead of 450 mg as per sponsor's decision, hence Cohort 2 and Cohort 3 have been combined.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Participants
  Non-SAE (>=5%) | 5 | 6 | 2 | 3 | 0
  SAE | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Amino Transferase (AST), Creatine Kinase (CK), Gamma-glutamyl Transferase (GGT) and Lactate Dehydrogenase (LDH) Over Time
Description: Blood samples were collected for the analysis of clinical parameters including ALT, ALP, CK, GGT, LDH and AST. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Days 29, 57, 85, 211
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles). In Cohort 3 participants were administered GSK3228836 300 mg instead of 450 mg as per sponsor's decision, hence Cohort 2 and Cohort 3 have been combined.
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Units per liter (U/L)
  ALT, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  ALT, Day29, n= 6,12,6,4,2 | 15.7 (56.65) | 52.5 (112.14) | -0.7 (8.91) | 45.3 (32.10) | -0.5 (3.54)
  ALT, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  ALT, Day57, n= 5,12,6,4,2 | 45.6 (60.06) | 37.5 (58.31) | -2.2 (8.77) | 46.0 (42.31) | 1.0 (3.54)
  ALT, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  ALT, Day85, n= 6,12,6,4,2 | -10.5 (30.20) | 8.8 (29.87) | 0.5 (9.14) | 7.5 (13.18) | -0.5 (0.71)
  ALT, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  ALT, Day211, n= 6,12,6,4,2 | -24.3 (43.68) | -16.2 (30.75) | -3.2 (12.88) | 6.5 (9.95) | 5.5 (3.54)
  ALP, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  ALP, Day29, n= 6,12,6,4,2 | -3.2 (8.23) | 5.2 (14.60) | -0.7 (8.12) | 9.8 (11.95) | 0.0 (0.90)
  ALP, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  ALP, Day57, n= 5,12,6,4,2 | 7.8 (12.09) | 13.3 (14.55) | 8.0 (11.31) | 1.3 (9.22) | 4.0 (5.66)
  ALP, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  ALP, Day85, n= 6,12,6,4,2 | 7.2 (7.73) | 9.9 (9.24) | 7.7 (9.89) | 0.0 (4.24) | 6.0 (4.24)
  ALP, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  ALP, Day211, n= 6,12,6,4,2 | 18.2 (10.32) | 11.3 (13.61) | 9.3 (8.71) | 1.5 (7.85) | 5.0 (11.31)
  AST, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  AST, Day29, n= 6,12,6,4,2 | 17.7 (50.41) | 31.0 (78.95) | -0.5 (3.99) | 27.5 (23.07) | 2.0 (1.41)
  AST, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  AST, Day57, n= 5,12,6,4,2 | 22.8 (34.30) | 23.3 (50.25) | 2.3 (3.33) | 18.3 (15.84) | 4.5 (2.12)
  AST, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  AST, Day85, n= 6,12,6,4,2 | 3.0 (16.66) | 4.6 (20.37) | 1.5 (4.46) | 5.5 (4.51) | 3.0 (0.00)
  AST, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  AST, Day211, n= 6,12,6,4,2 | -9.3 (22.20) | -6.5 (16.46) | 3.8 (3.76) | 5.3 (3.30) | 4.5 (2.12)
  CK, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  CK, Day29, n= 6,12,6,4,2 | 35.5 (127.87) | -17.6 (28.46) | -13.2 (29.36) | -6.8 (19.21) | 49.0 (62.23)
  CK, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  CK, Day57, n= 5,12,6,4,2 | -9.6 (47.77) | 9.8 (25.89) | -0.5 (24.04) | 57.0 (142.54) | 111.0 (148.49)
  CK, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  CK, Day85, n= 6,12,6,4,2 | 26.2 (61.64) | 16.8 (28.51) | 5.0 (49.78) | 178.8 (359.38) | 26.5 (31.82)
  CK, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  CK, Day211, n= 6,12,6,4,2 | 29.2 (71.04) | 24.2 (42.39) | 77.2 (132.59) | 53.8 (50.68) | 94.0 (114.55)
  GGT, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  GGT, Day29, n= 6,12,6,4,2 | -2.3 (3.88) | 3.1 (8.27) | -11.7 (22.27) | 5.3 (6.70) | -2.5 (2.12)
  GGT, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  GGT, Day57, n= 5,12,6,4,2 | 1.4 (3.44) | 6.5 (15.85) | -17.0 (36.30) | 9.0 (3.74) | 2.0 (2.83)
  GGT, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  GGT, Day85, n= 6,12,6,4,2 | -0.5 (1.52) | 3.2 (6.66) | -17.5 (37.56) | 5.3 (3.10) | 1.0 (2.83)
  GGT, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  GGT, Day211, n= 6,12,6,4,2 | -7.7 (11.57) | -1.1 (2.15) | -17.8 (41.06) | 4.3 (2.22) | 2.0 (1.41)
  LDH, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  LDH, Day29, n= 6,12,6,4,2 | 12.0 (27.03) | 1.7 (41.09) | -1.5 (15.00) | 46.8 (35.51) | 12.5 (0.71)
  LDH, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  LDH, Day57, n= 5,12,6,4,2 | 4.4 (26.68) | -4.7 (21.40) | 22.0 (36.74) | 4.8 (9.25) | 11.0 (11.31)
  LDH, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  LDH, Day85, n= 6,12,6,4,2 | 9.5 (22.79) | -12.3 (22.42) | 29.2 (35.29) | 3.8 (17.19) | 6.0 (8.49)
  LDH, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  LDH, Day211, n= 6,12,6,4,2 | 7.0 (18.78) | 3.3 (28.06) | 55.0 (54.59) | 25.3 (13.60) | 24.0 (22.63)

3. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters : Albumin and Total Protein Over Time
Description: Blood samples were collected for the analysis of clinical chemistry parameter-albumin and total protein. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Days 29, 57, 85, 211
Population: Safety population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). In Cohort 3 participants were administered GSK3228836 300 mg instead of 450 mg as per sponsor's decision, hence Cohort 2 and Cohort 3 have been combined.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Grams per liter
  Albumin, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Albumin, Day29, n= 6,12,6,4,2 | -0.8 (1.47) | 0.3 (2.23) | -1.3 (1.51) | 3.0 (2.16) | 1.5 (3.54)
  Albumin, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Albumin, Day57, n= 5,12,6,4,2 | 0.6 (1.67) | 1.7 (2.57) | 0.0 (1.55) | 1.8 (1.50) | 5.5 (0.71)
  Albumin, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Albumin, Day85, n= 6,12,6,4,2 | 0.0 (2.00) | 2.0 (3.28) | -0.8 (3.19) | 1.3 (2.22) | 3.0 (2.83)
  Albumin, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Albumin, Day211, n= 6,12,6,4,2 | 1.0 (2.28) | 3.3 (2.26) | 0.7 (3.01) | 4.3 (0.50) | 3.0 (5.66)
  Total Protein, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Total Protein, Day29, n= 6,12,6,4,2 | -1.8 (2.64) | 1.9 (3.18) | -1.8 (4.75) | 6.5 (3.11) | 1.5 (7.78)
  Total Protein, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Total Protein, Day57, n= 5,12,6,4,2 | 0.8 (3.49) | 3.8 (4.27) | 0.2 (3.25) | 3.0 (1.41) | 6.0 (0.0)
  Total Protein, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Total Protein, Day85, n= 6,12,6,4,2 | 0.8 (3.54) | 3.3 (5.03) | 0.3 (4.97) | 3.5 (3.42) | 4.5 (2.12)
  Total Protein, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Total Protein, Day211, n= 6,12,6,4,2 | 2.5 (4.81) | 5.1 (4.23) | 1.7 (3.33) | 8.0 (2.71) | 4.5 (12.02)

4. Primary Outcome: Change From Baseline Values in Clinical Chemistry Parameters: Sodium, Potassium, Chloride, Bicarbonate, Calcium, Magnesium, Phosphate, Glucose, Blood Urea Nitrogen, Cholesterol and Urate
Description: Blood samples were collected for the analysis of clinical parameters including sodium, potassium, chloride, bicarbonate, calcium, magnesium, phosphate, glucose, blood urea nitrogen (BUN), cholesterol and urate. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Outcome Measure Timeframe: Baseline (Day 1 pre-dose) and Days 29, 57, 85, 211
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Millimoles per liter
  Bicarbonate, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Bicarbonate, Day29, n= 6,12,6,4,2 | 0.3 (1.21) | 0.2 (1.11) | 1.0 (1.41) | 0.0 (2.16) | -2.0 (2.83)
  Bicarbonate, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Bicarbonate, Day57, n= 5,12,6,4,2 | 1.0 (2.65) | -0.1 (2.02) | -0.2 (2.14) | 0.3 (2.87) | -3.0 (2.83)
  Bicarbonate, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Bicarbonate, Day85, n= 6,12,6,4,2 | 0.2 (3.92) | 0.5 (1.83) | -0.8 (0.75) | -0.8 (0.50) | -2.0 (2.83)
  Bicarbonate, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Bicarbonate, Day211, n= 6,12,6,4,2 | 2.8 (1.94) | -1.0 (1.81) | -0.8 (1.72) | -0.8 (2.22) | -2.0 (4.24)
  Calcium, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Calcium, Day29, n= 6,12,6,4,2 | 0.012 (0.0811) | 0.015 (0.0735) | -0.040 (0.0506) | 0.063 (0.0479) | -0.030 (0.0707)
  Calcium, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Calcium, Day57, n= 5,12,6,4,2 | 0.036 (0.0658) | 0.029 (0.0899) | -0.038 (0.0471) | 0.013 (0.0150) | 0.010 (0.0566)
  Calcium, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Calcium, Day85, n= 6,12,6,4,2 | 0.020 (0.0672) | 0.046 (0.0944) | -0.028 (0.0679) | -0.013 (0.0675) | 0.050 (0.0707)
  Calcium, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Calcium, Day211, n= 6,12,6,4,2 | 0.052 (0.0618) | 0.056 (0.0745) | -0.025 (0.0789) | 0.068 (0.0746) | -0.025 (0.1344)
  Chloride, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Chloride, Day29, n= 6,12,6,4,2 | -0.8 (2.14) | -0.3 (1.97) | 0.8 (1.94) | -2.0 (1.83) | -1.5 (0.71)
  Chloride, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Chloride, Day57, n= 5,12,6,4,2 | -1.2 (2.17) | 0.0 (1.86) | 0.7 (0.82) | -1.0 (0.00) | -1.5 (0.71)
  Chloride, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Chloride, Day85, n= 6,12,6,4,2 | -1.0 (2.37) | 0.8 (1.85) | 1.5 (1.64) | -0.3 (1.50) | -1.5 (2.12)
  Chloride, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Chloride, Day211, n= 6,12,6,4,2 | -0.8 (2.48) | 0.0 (2.30) | 1.7 (2.94) | -0.5 (0.58) | -1.0 (1.41)
  Cholesterol, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Cholesterol, Day29, n= 6,12,6,4,2 | -0.027 (0.2281) | -0.129 (0.4305) | -0.252 (0.2044) | 0.123 (0.9238) | -0.155 (0.7000)
  Cholesterol, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Cholesterol, Day57, n= 5,12,6,4,2 | -0.422 (0.3739) | -0.328 (0.8109) | -0.717 (0.5216) | 0.480 (0.7278) | 0.815 (0.5303)
  Cholesterol, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Cholesterol, Day85, n= 6,12,6,4,2 | -0.380 (0.5772) | -0.211 (0.8659) | -0.812 (0.2704) | 0.195 (0.5073) | 0.390 (0.5091)
  Cholesterol, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Cholesterol, Day211, n= 6,12,6,4,2 | -0.110 (0.4369) | -0.121 (0.7581) | -0.423 (0.6980) | 0.960 (0.3982) | 0.360 (0.7354)
  Glucose, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Glucose, Day29, n= 6,12,6,4,2 | 0.170 (0.7148) | 0.009 (0.7782) | 0.498 (1.3437) | -0.290 (0.1299) | 0.225 (0.0778)
  Glucose, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Glucose, Day57, n= 5,12,6,4,2 | 0.056 (0.4161) | -0.110 (1.0510) | -0.157 (0.5147) | 0.415 (1.4055) | -0.360 (0.1980)
  Glucose, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Glucose, Day85, n= 6,12,6,4,2 | 0.018 (0.3725) | -0.218 (1.0970) | -0.315 (0.2959) | 0.073 (0.4524) | -0.110 (0.0000)
  Glucose, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Glucose, Day211, n= 6,12,6,4,2 | 0.093 (0.4956) | -0.205 (1.0796) | -0.223 (0.5205) | -0.373 (0.6375) | -0.110 (0.3111)
  Magnesium, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Magnesium, Day29, n= 6,12,6,4,2 | -0.008 (0.0376) | 0.013 (0.0377) | -0.025 (0.0524) | 0.000 (0.0000) | 0.025 (0.0354)
  Magnesium, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Magnesium, Day57, n= 5,12,6,4,2 | 0.000 (0.0500) | 0.038 (0.0483) | -0.033 (0.0516) | 0.013 (0.0479) | 0.000 (0.0000)
  Magnesium, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Magnesium, Day85, n= 6,12,6,4,2 | -0.025 (0.0612) | 0.029 (0.0620) | -0.033 (0.0606) | -0.038 (0.0479) | 0.000 (0.0000)
  Magnesium, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Magnesium, Day211, n= 6,12,6,4,2 | 0.008 (0.0585) | 0.042 (0.0669) | -0.008 (0.0492) | 0.050 (0.0577) | 0.025 (0.0354)
  Phosphate, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Phosphate, Day29, n= 6,12,6,4,2 | 0.052 (0.1488) | -0.010 (0.1123) | 0.023 (0.1472) | -0.073 (0.0562) | -0.050 (0.1131)
  Phosphate, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Phosphate, Day57, n= 5,12,6,4,2 | 0.052 (0.1657) | -0.064 (0.1072) | -0.025 (0.1088) | -0.058 (0.1250) | -0.020 (0.1556)
  Phosphate, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Phosphate, Day85, n= 6,12,6,4,2 | -0.020 (0.1942) | -0.003 (0.1342) | 0.055 (0.1001) | -0.008 (0.2017) | 0.080 (0.2546)
  Phosphate, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Phosphate, Day211, n= 6,12,6,4,2 | 0.023 (0.0528) | 0.056 (0.1800) | 0.005 (0.1401) | -0.018 (0.1231) | -0.130 (0.1273)
  Potassium, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Potassium, Day29, n= 6,12,6,4,2 | 0.08 (0.248) | 0.16 (0.215) | 0.12 (0.458) | -0.05 (0.289) | 0.00 (0.141)
  Potassium, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Potassium, Day57, n= 5,12,6,4,2 | 0.08 (0.335) | 0.27 (0.161) | 0.08 (0.293) | 0.03 (0.206) | -0.05 (0.354)
  Potassium, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Potassium, Day85, n= 6,12,6,4,2 | 0.07 (0.151) | 0.37 (0.183) | 0.20 (0.210) | 0.00 (0.476) | 0.00 (0.566)
  Potassium, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Potassium, Day211, n= 6,12,6,4,2 | 0.03 (0.367) | 0.31 (0.284) | 0.30 (0.228) | 0.23 (0.299) | 0.05 (0.919)
  Sodium, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Sodium, Day29, n= 6,12,6,4,2 | 0.2 (0.75) | 0.2 (2.33) | 0.7 (2.42) | -1.0 (2.16) | -1.5 (0.71)
  Sodium, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Sodium, Day57, n= 5,12,6,4,2 | -1.0 (1.87) | -0.2 (2.21) | -0.2 (1.47) | -0.5 (1.29) | -1.0 (0.00)
  Sodium, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Sodium, Day85, n= 6,12,6,4,2 | -0.3 (2.16) | 0.5 (2.28) | 0.2 (1.72) | -0.8 (1.71) | -2.0 (1.41)
  Sodium, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Sodium, Day211, n= 6,12,6,4,2 | -0.5 (2.35) | -0.3 (1.96) | 0.2 (1.94) | 0.3 (0.50) | -1.0 (0.00)
  Urate, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Urate, Day29, n= 6,12,6,4,2 | 0.0310 (0.05007) | 0.0248 (0.04039) | -0.0127 (0.01127) | -0.0060 (0.02728) | 0.0355 (0.04172)
  Urate, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Urate, Day57, n= 5,12,6,4,2 | 0.0192 (0.03713) | 0.0119 (0.05856) | -0.0158 (0.02260) | -0.0043 (0.04377) | 0.0030 (0.00424)
  Urate, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Urate, Day85, n= 6,12,6,4,2 | 0.0168 (0.04298) | -0.0061 (0.04391) | -0.0100 (0.02592) | -0.0078 (0.04984) | 0.0440 (0.02121)
  Urate, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Urate, Day211, n= 6,12,6,4,2 | 0.0012 (0.03783) | -0.0005 (0.05949) | -0.0128 (0.04086) | 0.0370 (0.02599) | 0.0325 (0.02899)
  BUN, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  BUN, Day29, n= 6,12,6,4,2 | 0.417 (1.0192) | 0.356 (0.5040) | 0.415 (0.6125) | 0.180 (0.8980) | 0.355 (1.0112)
  BUN, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  BUN, Day57, n= 5,12,6,4,2 | 0.788 (0.9903) | 0.238 (0.7960) | 0.535 (1.1451) | 0.980 (1.5543) | 0.180 (0.2546)
  BUN, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  BUN, Day85, n= 6,12,6,4,2 | -0.177 (0.9241) | -0.059 (0.8974) | 0.833 (0.7011) | 0.000 (1.2040) | 0.000 (0.5091)
  BUN, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  BUN, Day211, n= 6,12,6,4,2 | 0.358 (1.2580) | -0.208 (1.0941) | 0.713 (1.1510) | 0.893 (1.4463) | 0.000 (0.0000)

5. Primary Outcome: Change From Baseline Values in Clinical Chemistry Parameters: Total Bilirubin, Direct Bilirubin, Indirect Bilirubin, and Creatinine
Description: Blood samples were collected for the analysis of clinical chemistry parameters: direct bilirubin, total bilirubin, indirect bilirubin and creatinine. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Days 29, 57, 85, 211
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Micromoles per liter
  Total Bilirubin, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Total Bilirubin, Day29, n= 6,12,6,4,2 | -1.72 (2.699) | -1.07 (2.529) | -1.92 (2.497) | -1.53 (3.497) | 1.40 (1.414)
  Total Bilirubin, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Total Bilirubin, Day57, n= 5,12,6,4,2 | -2.14 (2.105) | -0.40 (3.930) | -1.72 (1.216) | -0.33 (3.802) | 3.85 (6.576)
  Total Bilirubin, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Total Bilirubin, Day85, n= 6,12,6,4,2 | -1.47 (2.151) | -0.78 (2.840) | -1.52 (3.411) | -0.78 (2.290) | 5.40 (7.071)
  Total Bilirubin, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Total Bilirubin, Day211, n= 6,12,6,4,2 | -0.87 (2.608) | -0.87 (3.538) | 0.40 (5.907) | 1.00 (2.432) | 2.75 (4.738)
  Direct Bilirubin, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Direct Bilirubin, Day29, n= 6,12,6,4,2 | 0.00 (0.000) | -0.02 (0.061) | 0.02 (0.041) | 0.00 (0.000) | 0.00 (0.000)
  Direct Bilirubin, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Direct Bilirubin, Day57, n= 5,12,6,4,2 | 0.00 (0.000) | -0.02 (0.061) | -0.07 (0.167) | 0.05 (0.105) | 0.00 (0.000)
  Direct Bilirubin, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Direct Bilirubin, Day85, n= 6,12,6,4,2 | 0.00 (0.000) | -0.02 (0.061) | -0.07 (0.167) | 0.00 (0.000) | 0.00 (0.000)
  Direct Bilirubin, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Direct Bilirubin, Day211, n= 6,12,6,4,2 | 0.00 (0.000) | -0.02 (0.061) | 0.05 (0.122) | 0.00 (0.000) | 0.00 (0.000)
  Indirect Bilirubin, Day29, n= 0,0,1,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Indirect Bilirubin, Day29, n= 0,0,1,0,0 |  |  | -0.60 (NA) — NA indicates that standard deviation could not be calculated for a single participant. |  |
  Indirect Bilirubin, Day57, n= 0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Indirect Bilirubin, Day85, n= 0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Indirect Bilirubin, Day211, n= 0,0,1,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Indirect Bilirubin, Day211, n= 0,0,1,0,0 |  |  | 10.50 (NA) — NA indicates that standard deviation could not be calculated for a single participant. |  |
  Creatinine, Day29, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Creatinine, Day29, n= 6,12,6,4,2 | 3.8 (3.39) | 7.8 (4.37) | -0.3 (7.00) | 8.8 (5.89) | 2.3 (3.18)
  Creatinine, Day57, n= 5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Creatinine, Day57, n= 5,12,6,4,2 | 2.7 (5.13) | 5.5 (6.53) | 2.5 (5.08) | 2.3 (12.18) | 2.3 (9.55)
  Creatinine, Day85, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Creatinine, Day85, n= 6,12,6,4,2 | 0.8 (8.73) | 3.9 (6.46) | 1.0 (5.67) | 2.0 (5.43) | 2.3 (3.18)
  Creatinine, Day211, n= 6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Creatinine, Day211, n= 6,12,6,4,2 | 0.8 (6.62) | 4.0 (8.82) | 4.0 (6.82) | 2.0 (5.43) | 6.8 (3.18)

6. Primary Outcome: Change From Baseline for Hematology Parameters: Basophils, Eosinophils, White Blood Cells (WBC), Lymphocytes, Neutrophils, Monocytes, and Platelets
Description: Blood samples were collected for the analysis of hematology parameters including basophil, eosinophils, WBC, lymphocytes, neutrophils, monocytes, and platelets at indicated timepoints. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Days 29, 57, 85, 211
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^9 cells per liters
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
10^9 cells per liters
  Basophils, Day 29: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Basophils, Day 29 | 0.00 (0.000) | 0.01 (0.029) | 0.00 (0.000) | 0.0 (0.00) | 0.0 (0.00)
  Basophils, Day 57: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Basophils, Day 57 | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.0 (0.00) | 0.0 (0.00)
  Basophils, Day 85: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Basophils, Day 85 | -0.02 (0.041) | 0.00 (0.000) | 0.00 (0.000) | 0.0 (0.00) | 0.0 (0.00)
  Basophils, Day 211: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Basophils, Day 211 | 0.00 (0.000) | 0.01 (0.029) | 0.00 (0.000) | 0.0 (0.00) | 0.0 (0.00)
  Eosinophils, Day 29: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Eosinophils, Day 29 | 0.03 (0.103) | -0.02 (0.103) | 0.03 (0.052) | 0.00 (0.082) | 0.00 (0.000)
  Eosinophils, Day 57: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Eosinophils, Day 57 | -0.02 (0.098) | -0.03 (0.115) | 0.05 (0.084) | 0.00 (0.082) | -0.10 (0.000)
  Eosinophils, Day 85: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Eosinophils, Day 85 | 0.08 (0.172) | -0.03 (0.115) | 0.02 (0.075) | -0.03 (0.126) | -0.05 (0.071)
  Eosinophils, Day 211: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Eosinophils, Day 211 | 0.10 (0.110) | -0.04 (0.108) | 0.03 (0.052) | 0.05 (0.058) | 0.05 (0.071)
  WBC, Day 29: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  WBC, Day 29 | -0.18 (1.206) | -0.60 (0.921) | -0.12 (0.826) | 0.28 (0.624) | -1.15 (0.212)
  WBC, Day 57: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  WBC, Day 57 | -0.33 (1.172) | -0.49 (0.958) | -0.37 (1.204) | 0.08 (0.222) | -0.95 (0.636)
  WBC, Day 85: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  WBC, Day 85 | -0.58 (1.177) | -0.63 (0.796) | -0.65 (0.814) | 0.43 (0.556) | -1.05 (0.071)
  WBC, Day 211: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  WBC, Day 211 | -0.45 (1.067) | 0.01 (0.696) | 0.10 (1.834) | 0.70 (0.589) | -0.85 (0.212)
  Lymphocytes, Day 29: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Lymphocytes, Day 29 | -0.10 (0.219) | -0.27 (0.293) | -0.03 (0.294) | -0.10 (0.216) | 0.20 (0.283)
  Lymphocytes Day 57: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Lymphocytes Day 57 | 0.00 (0.200) | -0.15 (0.275) | -0.10 (0.456) | -0.05 (0.100) | -0.05 (0.071)
  Lymphocytes, Day 85: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Lymphocytes, Day 85 | 0.17 (0.288) | -0.13 (0.273) | -0.03 (0.258) | 0.10 (0.294) | -0.10 (0.000)
  Lymphocytes, Day 211: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Lymphocytes, Day 211 | 0.17 (0.301) | -0.11 (0.334) | -0.07 (0.234) | 0.15 (0.208) | -0.10 (0.141)
  Neutrophils, Day 29: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Neutrophils, Day 29 | -0.17 (1.027) | -0.36 (0.945) | -0.17 (0.706) | 0.30 (0.392) | -1.05 (0.212)
  Neutrophils, Day 57: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Neutrophils, Day 57 | -0.30 (1.075) | -0.31 (0.898) | -0.32 (1.301) | 0.13 (0.275) | -0.60 (0.849)
  Neutrophils, Day 85: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Neutrophils, Day 85 | -0.95 (0.812) | -0.45 (1.026) | -0.67 (0.585) | 0.35 (0.342) | -0.65 (0.212)
  Neutrophils, Day 211: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Neutrophils, Day 211 | -0.75 (0.873) | 0.18 (0.725) | 0.08 (1.967) | 0.48 (0.377) | -0.55 (0.212)
  Monocytes, Day 29: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Monocytes, Day 29 | 0.08 (0.117) | -0.01 (0.138) | 0.02 (0.098) | 0.08 (0.050) | -0.25 (0.212)
  Monocytes, Day 57: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Monocytes, Day 57 | 0.00 (0.089) | -0.01 (0.131) | 0.00 (0.167) | 0.03 (0.096) | -0.15 (0.354)
  Monocytes, Day 85: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Monocytes, Day 85 | 0.08 (0.075) | -0.04 (0.124) | 0.03 (0.082) | 0.03 (0.050) | -0.20 (0.283)
  Monocytes, Day 211: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Monocytes, Day 211 | 0.07 (0.103) | -0.05 (0.100) | 0.02 (0.075) | 0.10 (0.115) | -0.15 (0.212)
  Platelets, Day 29: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Platelets, Day 29 | -0.5 (23.87) | -8.3 (17.23) | 11.0 (21.94) | 18.0 (32.28) | 16.0 (9.90)
  Platelets, Day 57: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Platelets, Day 57 | -2.5 (26.76) | -8.3 (31.77) | 9.7 (37.08) | -7.5 (8.70) | 24.5 (17.68)
  Platelets, Day 85: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Platelets, Day 85 | -5.2 (31.92) | -8.3 (29.59) | 22.2 (27.95) | 1.5 (7.14) | 14.5 (40.31)
  Platelets, Day 211: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Platelets, Day 211 | 12.3 (22.81) | 4.6 (43.15) | 25.8 (20.49) | 17.3 (20.52) | -4.5 (44.55)

7. Primary Outcome: Change From Baseline for Hematology Parameters: Hemoglobin
Description: Blood samples were collected for the analysis of hematology parameters including hemoglobin at indicated timepoints. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Days 29, 57, 85, 211
Population: Safety population. Only those participants with data available at the specified data points were analyzed. In Cohort 3 participants were administered GSK3228836 300 mg instead of 450 mg as per sponsor's decision, hence Cohort 2 and Cohort 3 have been combined.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
Grams per liter
  Day 29 | -7.3 (3.50) | -6.8 (8.74) | -11.3 (7.31) | -6.0 (6.48) | -11.5 (2.12)
  Day 57 | -3.3 (10.25) | -3.0 (10.79) | -5.8 (9.28) | -3.8 (6.95) | -3.5 (4.95)
  Day 85 | -4.0 (10.60) | -4.8 (13.13) | -9.2 (10.07) | -0.3 (3.86) | -5.0 (9.90)
  Day 211 | -0.7 (15.73) | 1.8 (16.68) | -7.5 (6.47) | 4.8 (5.19) | 0.0 (1.41)

8. Primary Outcome: Change From Baseline for Hematology Parameter: Hematocrit
Description: Blood samples were collected for the analysis of hematology parameter including hematocrit at indicated timepoints. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Days 29, 57, 85, 211
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
Percentage of red blood cells in blood
  Day 29 | -2.47 (1.150) | -2.39 (2.858) | -4.20 (2.577) | -2.23 (2.089) | -3.30 (0.283)
  Day 57 | -1.17 (2.630) | -1.04 (3.089) | -2.17 (3.080) | -1.10 (2.482) | -0.80 (2.546)
  Day 85 | -1.33 (3.043) | -0.98 (3.698) | -3.13 (2.501) | -0.28 (1.646) | -1.65 (3.748)
  Day 211 | -0.37 (4.065) | 1.53 (4.799) | -1.83 (2.066) | 1.40 (1.930) | 1.05 (1.768)

9. Primary Outcome: Change From Baseline Values in Urine Specific Gravity
Description: Urine samples were collected for the analysis of urine specific gravity. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value. Urine specific gravity is measured as the ratio of urine density compared with water density.
Time Frame: Baseline (Day 1 pre-dose) and Days 29, 57, 85, 211
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Ratio of urine to water density
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
Ratio of urine to water density
  Day 29 | -0.0017 (0.00703) | 0.0033 (0.00585) | 0.0032 (0.00523) | 0.0028 (0.00427) | 0.0080 (0.00566)
  Day 57 | 0.0000 (0.00832) | 0.0059 (0.00763) | 0.0028 (0.00519) | 0.0038 (0.00457) | 0.0130 (0.00141)
  Day 85 | -0.0007 (0.00653) | 0.0020 (0.00481) | 0.0057 (0.00441) | 0.0013 (0.00450) | 0.0130 (0.00000)
  Day 211 | -0.0020 (0.00851) | 0.0024 (0.00684) | 0.0010 (0.00522) | -0.0005 (0.00387) | 0.0060 (0.00849)

10. Primary Outcome: Change From Baseline Values in Urine Albumin/Creatinine Ratio and Urine Protein/Creatinine Ratio
Description: Urine samples were collected for the analysis of urine albumin/creatinine ratio and urine protein/creatinine ratio. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Days 29, 57, 85, 211
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Milligrams per millimole Creatinine
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Milligrams per millimole Creatinine
  Urine albumin/creatinine ratio, Day29,n=0,1,0,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Urine albumin/creatinine ratio, Day29,n=0,1,0,0,0 |  | -3.340 (NA) — NA indicates that standard deviation could not be calculated for a single participant. |  |  |
  Urine albumin/creatinine ratio, Day57,n=0,2,0,0,0: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0
  Urine albumin/creatinine ratio, Day57,n=0,2,0,0,0 |  | -10.580 (10.9743) |  |  |
  Urine albumin/creatinine ratio, Day85,n=0,1,1,0,0: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  Urine albumin/creatinine ratio, Day85,n=0,1,1,0,0 |  | -3.480 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 0.080 (NA) — NA indicates that standard deviation could not be calculated for a single participant. |  |
  Urine albumin/creatinine ratio, Day211,n=0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Urine protein/creatinine ratio Day29, n=5,10,4,4,2: number analyzed (Participants) | 5 | 10 | 4 | 4 | 2
  Urine protein/creatinine ratio Day29, n=5,10,4,4,2 | 0.006 (0.0329) | -0.002 (0.1264) | -0.005 (0.0058) | 0.065 (0.0238) | 0.025 (0.0071)
  Urine protein/creatinine ratio Day57, n=6,9,3,4,2: number analyzed (Participants) | 6 | 9 | 3 | 4 | 2
  Urine protein/creatinine ratio Day57, n=6,9,3,4,2 | -0.007 (0.0589) | -0.043 (0.1168) | -0.003 (0.0058) | 0.020 (0.0000) | 0.010 (0.0000)
  Urine protein/creatinine ratio Day85, n=6,8,4,3,2: number analyzed (Participants) | 6 | 8 | 4 | 3 | 2
  Urine protein/creatinine ratio Day85, n=6,8,4,3,2 | -0.003 (0.0554) | -0.050 (0.1042) | -0.005 (0.0129) | 0.017 (0.0231) | 0.000 (0.0141)
  Urine protein/creatinine ratio Day211, n=4,8,4,3,1: number analyzed (Participants) | 4 | 8 | 4 | 3 | 1
  Urine protein/creatinine ratio Day211, n=4,8,4,3,1 | 0.003 (0.0150) | -0.073 (0.1235) | -0.005 (0.0311) | 0.013 (0.0252) | 0.000 (NA) — NA indicates that standard deviation could not be calculated for a single participant.

11. Primary Outcome: Change From Baseline Values in Urine Protein
Description: Urine samples were collected for the analysis of urine protein. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Days 29, 57, 85, 211
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
Milligrams per deciliter
  Day 29 | -1.08 (7.591) | 7.06 (5.130) | -0.51 (2.605) | 11.13 (9.288) | 3.76 (5.020)
  Day 57 | -2.57 (7.451) | 5.62 (7.910) | 2.00 (5.903) | 4.48 (3.502) | 5.56 (3.889)
  Day 85 | -2.07 (5.814) | 1.45 (3.747) | 2.29 (2.267) | 2.48 (3.954) | 4.01 (0.283)
  Day 211 | -2.29 (7.277) | 0.90 (2.832) | -0.46 (2.214) | 0.90 (1.664) | 2.71 (3.8250)

12. Primary Outcome: Change From Baseline Values in Blood Coagulation Factors: Activated Partial Thromboplastin Time and Prothrombin Time
Description: Blood samples were collected for the analysis of blood coagulation factors:activated partial thromboplastin time (aPTT) and Prothrombin Time (PT). Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Days 23, 57, 85, 211
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Seconds
  aPTT, Day 23, n=5,11,6,4,2: number analyzed (Participants) | 5 | 11 | 6 | 4 | 2
  aPTT, Day 23, n=5,11,6,4,2 | -2.44 (4.017) | -2.33 (6.460) | -1.63 (1.715) | -0.45 (1.808) | 0.65 (0.778)
  aPTT, Day 57, n=6,12,5,4,2: number analyzed (Participants) | 6 | 12 | 5 | 4 | 2
  aPTT, Day 57, n=6,12,5,4,2 | 1.23 (3.518) | -3.03 (5.854) | -0.18 (3.841) | 0.13 (3.627) | -0.35 (1.344)
  aPTT, Day 85, n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  aPTT, Day 85, n=0,0,0,1,0 |  |  |  | 0.00 (NA) — NA indicates that standard deviation could not be calculated for a single participant. |
  aPTT, Day 211, n=5,11,6,2,2: number analyzed (Participants) | 5 | 11 | 6 | 2 | 2
  aPTT, Day 211, n=5,11,6,2,2 | 1.28 (6.538) | -1.01 (6.310) | 2.70 (3.046) | 1.30 (4.384) | 2.60 (3.394)
  PT, Day 23, n=5,11,6,4,2: number analyzed (Participants) | 5 | 11 | 6 | 4 | 2
  PT, Day 23, n=5,11,6,4,2 | -0.42 (0.576) | -0.23 (0.710) | 0.12 (0.483) | 0.33 (0.585) | 0.60 (0.141)
  PT, Day 57, n=6,12,5,4,2: number analyzed (Participants) | 6 | 12 | 5 | 4 | 2
  PT, Day 57, n=6,12,5,4,2 | -0.10 (0.740) | -0.50 (0.615) | 0.20 (0.869) | -0.18 (0.780) | 0.40 (0.141)
  PT, Day85, n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  PT, Day85, n=0,0,0,1,0 |  |  |  | -0.80 (NA) — NA indicates that standard deviation could not be calculated for a single participant. |
  PT, Day211, n=5,11,6,2,2: number analyzed (Participants) | 5 | 11 | 6 | 2 | 2
  PT, Day211, n=5,11,6,2,2 | -0.84 (0.623) | -0.35 (0.726) | 0.42 (0.744) | 0.45 (0.919) | 0.70 (0.283)

13. Primary Outcome: Change From Baseline Values in Blood Coagulation Factor: Prothrombin International Normalized Ratio
Description: Blood samples were collected for the analysis of blood coagulation factor: Prothrombin International normalized ratio. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Days 23, 57, 85, 211
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Ratio
  Day 23, n=5,11,6,4,2: number analyzed (Participants) | 5 | 11 | 6 | 4 | 2
  Day 23, n=5,11,6,4,2 | -0.04 (0.055) | -0.04 (0.067) | 0.02 (0.041) | 0.03 (0.096) | 0.00 (0.000)
  Day 57, n=6,12,5,4,2: number analyzed (Participants) | 6 | 12 | 5 | 4 | 2
  Day 57, n=6,12,5,4,2 | -0.02 (0.075) | -0.04 (0.079) | 0.02 (0.084) | 0.00 (0.082) | 0.00 (0.000)
  Day 85, n=0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Day 85, n=0,0,0,1,0 |  |  |  | 0.00 (NA) — NA indicates that standard deviation could not be calculated for a single participant. |
  Day 211, n=5,11,6,2,2: number analyzed (Participants) | 5 | 11 | 6 | 2 | 2
  Day 211, n=5,11,6,2,2 | -0.06 (0.089) | -0.03 (0.079) | 0.02 (0.075) | 0.05 (0.071) | 0.00 (0.000)

14. Primary Outcome: Change in Complement C3 Level at Worst Case Post Baseline Relative to Baseline
Description: Blood samples were collected from participants to evaluate change in complement C3 level at worst case post Baseline relative to Baseline. Worst case post Baseline in Complement C3 was the minimum post-Baseline level. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and up to Day 211
Population: Safety Population. In Cohort 3 participants were administered GSK3228836 300 mg instead of 450 mg as per sponsor's decision, hence Cohort 2 and Cohort 3 have been combined.
Measure: Mean (Standard Deviation); unit: Milligram per deciliter
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Milligram per deciliter | -19.8 (11.72) | -22.3 (12.00) | -16.5 (13.81) | -12.4 (3.78) | -25.5 (16.26)

15. Primary Outcome: Change in Complement C5a Level at Worst Case Post Baseline Relative to Baseline
Description: Blood samples were collected from participants to evaluate change in complement C5a level at worst case post Baseline relative to Baseline. Worst case post Baseline in Complement C5a was the maximum post-Baseline level. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and up to Day 211
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Nanogram per milliliter | 1.552 (1.3967) | 3.778 (6.2062) | 1.303 (0.8671) | 2.232 (2.2640) | 0.800 (0.0000)

16. Primary Outcome: Change in Complement Bb Level at Worst Case Post Baseline Relative to Baseline
Description: Blood samples were collected from participants to evaluate change in complement Bb level at worst case post Baseline relative to Baseline. Worst case post Baseline in Complement Bb was the maximum post-Baseline level. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and up to Day 211
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Microgram per milliliter | 0.355 (0.1129) | 0.365 (0.4835) | 0.240 (0.3543) | 0.472 (0.1439) | 0.320 (0.3677)

17. Primary Outcome: Number of Participants With Reported Pregnancy
Description: Female participants who were not surgically sterile or post-menopausal, underwent urine beta Human chorionic gonadotropin (Beta-HCG) pregnancy test.
Time Frame: Up to Day 211
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 3 | 8 | 2 | 1 | 1
Participants | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Change From Baseline in Body Temperature
Description: Body temperature was measured at indicated timepoints. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Days 29, 57, 85, 211
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
Degrees Celsius
  Day 29 | -0.05 (0.288) | -0.09 (0.353) | -0.15 (0.164) | 0.08 (0.250) | 0.30 (0.141)
  Day 57 | 0.03 (0.294) | -0.16 (0.342) | -0.18 (0.248) | 0.48 (0.096) | 0.20 (0.849)
  Day 85 | 0.05 (0.451) | -0.18 (0.290) | -0.13 (0.103) | 0.10 (0.115) | -0.20 (0.707)
  Day 211 | -0.20 (0.210) | -0.19 (0.291) | -0.17 (0.216) | 0.23 (0.369) | -0.10 (0.424)

19. Primary Outcome: Change From Baseline in Body Weight
Description: Body weight was measured at indicated time points. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Days 29, 57, 211
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
Kilograms
  Day 29 | -0.48 (3.406) | 0.20 (0.802) | 0.52 (0.786) | 0.00 (0.808) | -1.25 (0.636)
  Day 57 | -0.40 (3.992) | -0.10 (1.834) | -0.18 (1.009) | 0.20 (1.214) | -0.25 (0.354)
  Day 211 | -0.15 (3.627) | -0.40 (2.721) | -0.37 (1.350) | 2.00 (1.212) | 1.95 (0.354)

20. Primary Outcome: Change From Baseline in Diastolic Blood Pressure and Systolic Blood Pressure
Description: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP) was measured at indicated timepoints. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Days 29, 57, 85, 211
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
Millimeters of Mercury (mmHg)
  SBP, Day 29 | -6.3 (13.76) | -8.8 (12.05) | -9.2 (10.11) | -3.0 (6.63) | 0.5 (9.19)
  SBP, Day 57 | 3.7 (11.33) | -3.4 (13.98) | -13.2 (5.31) | 7.8 (7.93) | -2.0 (5.66)
  SBP, Day 85 | 3.0 (12.44) | -5.4 (13.45) | -13.7 (7.99) | 4.3 (8.58) | 6.5 (13.44)
  SBP, Day 211 | 10.0 (13.49) | -3.6 (15.21) | -10.2 (5.19) | 7.3 (10.21) | 5.0 (9.90)
  DBP, Day 29 | -4.0 (8.65) | -2.2 (7.77) | -6.0 (5.73) | -5.0 (7.26) | -0.5 (9.19)
  DBP, Day 57 | 1.0 (8.20) | -0.2 (9.92) | -3.0 (11.06) | 0.0 (9.38) | 3.0 (4.24)
  DBP, Day 85 | 2.2 (6.71) | 0.1 (12.43) | -3.7 (6.65) | -1.8 (6.08) | 4.5 (14.85)
  DBP, Day 211 | 6.8 (6.37) | 0.8 (9.88) | -3.8 (9.56) | 4.3 (6.95) | 8.0 (8.49)

21. Primary Outcome: Change From Baseline in Respiratory Rate
Description: Respiratory Rate was measured at indicated timepoints. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Days 29, 57, 85, 211
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Breaths/minute
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
Breaths/minute
  Day 29 | 0.3 (1.03) | 0.7 (0.65) | 0.3 (0.52) | -0.8 (2.22) | -2.5 (2.12)
  Day 57 | -0.5 (1.87) | 0.6 (0.67) | 0.2 (1.33) | -0.8 (2.22) | -2.5 (2.12)
  Day 85 | -0.3 (1.86) | 0.5 (0.52) | 0.2 (0.41) | -0.8 (2.22) | -3.0 (1.41)
  Day 211 | -0.5 (1.97) | 0.7 (0.78) | 0.0 (0.10) | -1.0 (2.00) | -3.0 (1.41)

22. Primary Outcome: Change From Baseline in Pulse Rate
Description: Pulse Rate was measured at indicated timepoints. Baseline value is defined as last non-missing measurement prior to the first dose of study drug. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Days 29, 57, 85, 211
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
Beats/minute
  Day 29 | -4.7 (13.63) | 4.3 (8.14) | 1.5 (5.32) | 9.0 (6.63) | 1.0 (4.24)
  Day 57 | -1.5 (16.34) | 8.2 (14.33) | 6.5 (14.36) | 16.0 (6.06) | 8.0 (4.24)
  Day 85 | 5.7 (19.96) | 2.3 (9.10) | -1.7 (7.15) | 16.8 (5.32) | 3.5 (7.78)
  Day 211 | -0.3 (18.82) | 2.9 (8.70) | 1.8 (12.22) | 16.3 (8.42) | 13.0 (2.83)

23. Primary Outcome: Number of Participants With Abnormal Findings in Physical Examination
Description: Physical examinations included assessment of the dermatologic, cardiovascular, respiratory, gastrointestinal, and neurological systems.
Time Frame: Up to Day 211
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Participants | 3 | 1 | 1 | 0 | 0

24. Primary Outcome: Number of Participants Who Received Atleast One Concomitant Medication
Description: A concomitant medication is defined as any medication initiated after the first dose of study, or initiated prior to the first dose of study drug and continued after the first dose of study drug.
Time Frame: Up to Day 211
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Participants | 4 | 8 | 5 | 5 | 2

25. Primary Outcome: Change From Baseline in Electrocardiogram Mean Ventricular Rate
Description: Triplicate 12-lead Electrocardiograms (ECGs) were recorded at indicated timepoints. At each time point, ECG machine automatically measured mean ventricular rate (VR). Baseline ECG was the average of the triplicate taken on Day 1 Pre-dose, if only 1 or 2 assessments were available, the single assessment or average of the 2 assessments was used. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose); Day1: 3 hours post-dose, 5 hours post-dose; Day 2; Day 22:pre-dose, 3 hours postdose, 5 hours post-dose; Days 23, 29 and 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Beats per minute
  Mean VR, Day1, 3 hours Post-dose, n=6,12,6,5,2 | 4.3 (5.05) | 5.6 (8.85) | 4.5 (4.93) | 8.2 (4.60) | 10.0 (2.83)
  Mean VR, Day1, 5 hours Post-dose, n=6,12,6,5,2 | 1.8 (6.52) | 2.0 (7.93) | 4.7 (6.22) | 12.6 (6.88) | 8.0 (9.90)
  Mean VR, Day 2, n=6,12,6,5,2 | -2.7 (10.27) | 10.1 (12.93) | 0.3 (2.66) | 22.8 (9.15) | 5.5 (7.78)
  Mean VR, Day 22, Pre-dose, n=5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Mean VR, Day 22, Pre-dose, n=5,12,6,4,2 | -3.6 (5.46) | 0.4 (8.54) | 1.0 (6.54) | 0.8 (4.86) | -1.0 (5.66)
  Mean VR, Day 22, 3 hours Post-dose, n=5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Mean VR, Day 22, 3 hours Post-dose, n=5,12,6,4,2 | -1.4 (7.37) | 5.0 (7.24) | 3.7 (5.47) | 9.3 (4.92) | 8.5 (2.12)
  Mean VR, Day 22, 5 hours Post-dose, n=5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Mean VR, Day 22, 5 hours Post-dose, n=5,12,6,4,2 | -1.8 (10.47) | 3.4 (6.27) | -0.7 (5.82) | 8.0 (6.22) | 8.0 (2.83)
  Mean VR, Day 23, n=5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  Mean VR, Day 23, n=5,12,6,4,2 | -2.4 (8.26) | 6.3 (3.65) | 1.3 (4.76) | 10.3 (4.92) | 0.0 (4.24)
  Mean VR, Day 29, n=6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Mean VR, Day 29, n=6,12,6,4,2 | -1.3 (11.60) | 2.8 (7.63) | 0.2 (4.45) | 7.3 (6.13) | 3.5 (7.78)
  Mean VR, Day 113, n=6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  Mean VR, Day 113, n=6,12,6,4,2 | -5.2 (9.75) | 2.5 (10.60) | -2.3 (6.06) | 8.3 (2.06) | 8.0 (9.90)

26. Primary Outcome: Change From Baseline in PR Interval, QRS Duration, Uncorrected QT Interval, QT Corrected Interval-Fredericia Interval and QTc Corrected by Bazett's Formula
Description: Triplicate 12-lead Electrocardiograms (ECGs) were recorded at indicated timepoints. At each time point, ECG machine automatically measured QRS duration, uncorrected QT interval, QT corrected interval-Fredericia [QTcF] interval and QTc corrected by Bazett's formula (QTcB). Baseline ECG was the average of the triplicate taken on Day 1 Pre-dose, if only 1 or 2 assessments were available, the single assessment or average of the 2 assessments was used. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: as for outcome 25
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Milliseconds
  PR, Day 1,3 hours Post-dose, n=6,11,6,5,2: number analyzed (Participants) | 6 | 11 | 6 | 5 | 2
  PR, Day 1,3 hours Post-dose, n=6,11,6,5,2 | -1.2 (8.42) | 1.8 (9.99) | 3.5 (30.84) | 0.8 (8.41) | 7.0 (1.41)
  PR, Day 1, 5 hours Post-dose, n=6,11,6,5,2: number analyzed (Participants) | 6 | 11 | 6 | 5 | 2
  PR, Day 1, 5 hours Post-dose, n=6,11,6,5,2 | -1.7 (8.64) | 1.3 (8.37) | 10.8 (33.52) | 1.4 (8.38) | -3.0 (0.00)
  PR, Day 2, n=6,12,6,5,2 | 1.0 (4.65) | 0.7 (15.78) | 12.2 (21.45) | -2.4 (8.79) | 5.5 (2.12)
  PR, Day 22, Pre-dose, n=5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  PR, Day 22, Pre-dose, n=5,12,6,4,2 | 7.0 (14.27) | -2.4 (11.70) | 11.0 (19.84) | -2.8 (10.87) | 8.0 (7.07)
  PR, Day 22, 3 hours Post-dose, n=5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  PR, Day 22, 3 hours Post-dose, n=5,12,6,4,2 | 2.0 (7.21) | 0.3 (14.51) | 9.2 (21.51) | -6.5 (11.79) | 7.5 (6.36)
  PR, Day 22, 5 hours Post-dose, n=5,11,6,4,2: number analyzed (Participants) | 5 | 11 | 6 | 4 | 2
  PR, Day 22, 5 hours Post-dose, n=5,11,6,4,2 | -0.2 (10.03) | -2.3 (14.18) | 9.0 (22.82) | -7.0 (9.42) | 5.5 (4.95)
  PR, Day 23, n=5,11,6,4,2: number analyzed (Participants) | 5 | 11 | 6 | 4 | 2
  PR, Day 23, n=5,11,6,4,2 | 9.4 (12.03) | -1.6 (11.09) | 11.2 (21.77) | -1.0 (7.79) | 4.5 (3.54)
  PR, Day 29, n=6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  PR, Day 29, n=6,12,6,4,2 | 4.8 (7.28) | -1.7 (11.67) | 7.3 (17.64) | -1.8 (4.72) | 10.0 (4.24)
  PR, Day 113, n=6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  PR, Day 113, n=6,12,6,4,2 | 7.7 (8.82) | -1.6 (14.48) | 14.3 (21.81) | -2.0 (8.83) | 6.0 (7.07)
  QRS duration, Day1, 3 hours Post-dose,n=6,12,6,5,2 | 0.8 (3.97) | -0.2 (5.08) | 2.2 (4.31) | 1.0 (2.00) | -1.5 (3.54)
  QRS duration, Day1, 5 hours Post-dose,n=6,12,6,5,2 | -0.8 (2.04) | -1.7 (4.38) | 6.0 (4.98) | 0.4 (1.95) | -3.0 (4.24)
  QRS duration, Day 2, n=6,12,6,5,2 | 0.5 (3.94) | 0.8 (3.98) | 3.7 (8.07) | -2.2 (4.87) | -0.5 (0.71)
  QRS duration, Day 22, Pre-dose, n=5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  QRS duration, Day 22, Pre-dose, n=5,12,6,4,2 | 0.2 (3.11) | -3.6 (5.07) | 4.2 (3.19) | -0.8 (4.79) | -4.0 (2.83)
  QRS duration, Day 22, 3 hours Post-dose, n=5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  QRS duration, Day 22, 3 hours Post-dose, n=5,12,6,4,2 | 1.6 (3.51) | -1.2 (4.11) | 5.0 (6.99) | 2.5 (1.91) | -1.0 (0.00)
  QRS duration, Day 22, 5 hours Post-dose, n=5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  QRS duration, Day 22, 5 hours Post-dose, n=5,12,6,4,2 | 1.0 (5.15) | -1.0 (3.86) | 6.3 (5.28) | -0.3 (5.12) | -2.0 (1.41)
  QRS duration, Day 23, n=5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  QRS duration, Day 23, n=5,12,6,4,2 | -0.4 (5.37) | 0.9 (3.09) | 0.3 (7.00) | -0.5 (4.12) | 1.5 (3.54)
  QRS duration, Day 29, n=6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  QRS duration, Day 29, n=6,12,6,4,2 | 0.3 (4.18) | 0.7 (4.91) | 5.5 (7.50) | 3.0 (6.98) | 0.5 (0.71)
  QRS duration, Day 113, n=6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  QRS duration, Day 113, n=6,12,6,4,2 | 0.3 (5.72) | 0.0 (4.90) | 4.7 (8.09) | -2.8 (5.19) | 1.0 (1.41)
  QT, Day 1, 3 hours Post-dose, n=6,12,6,5,2 | -11.8 (14.85) | -12.4 (17.30) | -5.7 (8.21) | -23.8 (9.55) | -20.5 (0.71)
  QT, Day 1, 5 hours Post-dose, n=6,12,6,5,2 | -11.3 (19.41) | -10.3 (18.25) | -7.3 (12.80) | -37.6 (19.89) | -21.0 (11.31)
  QT, Day 2, n=6,12,6,5,2 | -0.3 (29.34) | -25.5 (29.57) | 0.3 (6.41) | -62.8 (19.38) | 19.5 (19.09)
  QT, Day 22, Pre-dose, n=5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  QT, Day 22, Pre-dose, n=5,12,6,4,2 | 15.2 (12.91) | 1.9 (17.05) | 2.0 (19.65) | -1.0 (12.68) | 3.0 (11.31)
  QT, Day 22, 3 hours Post-dose, n=5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  QT, Day 22, 3 hours Post-dose, n=5,12,6,4,2 | 11.2 (30.60) | -8.7 (21.05) | -3.0 (17.31) | -27.3 (22.47) | -16.0 (12.73)
  QT, Day 22, 5 hours Post-dose, n=5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  QT, Day 22, 5 hours Post-dose, n=5,12,6,4,2 | 5.8 (29.71) | -8.0 (18.68) | 2.5 (16.31) | -25.3 (23.73) | -17.5 (9.19)
  QT, Day 23, n=5,12,6,4,2: number analyzed (Participants) | 5 | 12 | 6 | 4 | 2
  QT, Day 23, n=5,12,6,4,2 | 8.0 (23.63) | -13.9 (13.81) | -5.2 (16.74) | -30.5 (18.81) | -8.5 (6.36)
  QT, Day 29, n=6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  QT, Day 29, n=6,12,6,4,2 | 9.0 (31.92) | -5.4 (20.97) | 2.5 (15.45) | -23.0 (16.02) | -4.0 (31.11)
  QT, Day 113, n=6,12,6,4,2: number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
  QT, Day 113, n=6,12,6,4,2 | 13.7 (30.59) | -15.4 (49.82) | 4.2 (17.95) | -28.3 (13.33) | -20.0 (22.63)
  QTcB, Day 1,3 hours Post-dose, n=1,3,2,0,0: number analyzed (Participants) | 1 | 3 | 2 | 0 | 0
  QTcB, Day 1,3 hours Post-dose, n=1,3,2,0,0 | 5.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 3.3 (3.06) | 3.0 (1.41) |  |
  QTcB, Day 1, 5 hours Post-dose, n=1,3,2,0,0: number analyzed (Participants) | 1 | 3 | 2 | 0 | 0
  QTcB, Day 1, 5 hours Post-dose, n=1,3,2,0,0 | -9.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | -1.3 (11.02) | 4.5 (0.71) |  |
  QTcB, Day 2, n=1,3,2,0,0: number analyzed (Participants) | 1 | 3 | 2 | 0 | 0
  QTcB, Day 2, n=1,3,2,0,0 | -3.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 4.3 (7.57) | 2.5 (0.71) |  |
  QTcB, Day 22, Pre-dose, n=1,3,2,0,0: number analyzed (Participants) | 1 | 3 | 2 | 0 | 0
  QTcB, Day 22, Pre-dose, n=1,3,2,0,0 | 27.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 7.3 (6.43) | -0.5 (7.78) |  |
  QTcB, Day 22, 3 hours Post-dose, n=1,3,2,0,0: number analyzed (Participants) | 1 | 3 | 2 | 0 | 0
  QTcB, Day 22, 3 hours Post-dose, n=1,3,2,0,0 | 16.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 18.7 (16.77) | -2.0 (2.83) |  |
  QTcB, Day 22, 5 hours Post-dose, n=1,3,2,0,0: number analyzed (Participants) | 1 | 3 | 2 | 0 | 0
  QTcB, Day 22, 5 hours Post-dose, n=1,3,2,0,0 | 11.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 3.7 (2.31) | -14.5 (6.36) |  |
  QTcB, Day 23, n=1,3,2,0,0: number analyzed (Participants) | 1 | 3 | 2 | 0 | 0
  QTcB, Day 23, n=1,3,2,0,0 | 14.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 7.3 (8.62) | -3.5 (7.78) |  |
  QTcB, Day 29, n=1,4,2,0,0: number analyzed (Participants) | 1 | 4 | 2 | 0 | 0
  QTcB, Day 29, n=1,4,2,0,0 | 21.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 3.0 (8.98) | 6.5 (6.36) |  |
  QTcB, Day 113, n=1,5,3,0,0: number analyzed (Participants) | 1 | 5 | 3 | 0 | 0
  QTcB, Day 113, n=1,5,3,0,0 | 5.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | -1.8 (3.27) | -13.0 (8.54) |  |
  QTcF, Day 1,3 hours Post-dose, n=5,9,4,5,2: number analyzed (Participants) | 5 | 9 | 4 | 5 | 2
  QTcF, Day 1,3 hours Post-dose, n=5,9,4,5,2 | -6.0 (6.28) | -1.9 (8.16) | 3.5 (7.05) | -3.8 (13.88) | -4.5 (4.95)
  QTcF, Day 1,5 hours Post-dose, n=5,9,4,5,2: number analyzed (Participants) | 5 | 9 | 4 | 5 | 2
  QTcF, Day 1,5 hours Post-dose, n=5,9,4,5,2 | -9.6 (10.67) | -8.9 (8.49) | 1.3 (5.32) | -9.0 (13.84) | -7.5 (6.36)
  QTcF, Day 2, n=4,8,4,5,2: number analyzed (Participants) | 4 | 8 | 4 | 5 | 2
  QTcF, Day 2, n=4,8,4,5,2 | -8.6 (13.50) | -12.5 (9.01) | -1.0 (4.69) | -44.6 (65.50) | -11.0 (5.66)
  QTcF, Day 22, Pre-dose, n=5,9,4,4,2: number analyzed (Participants) | 5 | 9 | 4 | 4 | 2
  QTcF, Day 22, Pre-dose, n=5,9,4,4,2 | -1.0 (2.94) | 0.7 (12.19) | 8.8 (8.88) | 1.3 (3.77) | -1.5 (2.12)
  QTcF, Day 22, 3 hours Post-dose, n=4,9,4,4,2: number analyzed (Participants) | 4 | 9 | 4 | 4 | 2
  QTcF, Day 22, 3 hours Post-dose, n=4,9,4,4,2 | 0.8 (10.08) | -1.0 (11.10) | 9.5 (10.47) | -4.5 (13.48) | -1.5 (10.61)
  QTcF, Day 22, 5 hours Post-dose, n=4,9,4,5,2: number analyzed (Participants) | 4 | 9 | 4 | 5 | 2
  QTcF, Day 22, 5 hours Post-dose, n=4,9,4,5,2 | -5.0 (7.66) | -3.6 (12.97) | 5.8 (9.95) | -5.8 (12.55) | -4.5 (4.95)
  QTcF, Day 23, n=4,8,4,4,2: number analyzed (Participants) | 4 | 8 | 4 | 4 | 2
  QTcF, Day 23, n=4,8,4,4,2 | -0.8 (8.38) | -3.3 (9.82) | -0.5 (7.05) | -5.0 (9.20) | -10.0 (0.00)
  QTcF, Day 29, n=5,8,4,4,2: number analyzed (Participants) | 5 | 8 | 4 | 4 | 2
  QTcF, Day 29, n=5,8,4,4,2 | 4.0 (22.55) | -0.1 (9.60) | 3.0 (8.98) | -5.5 (10.08) | -4.5 (10.61)
  QTcF, Day 113, n=5,6,3,4,2: number analyzed (Participants) | 5 | 6 | 3 | 4 | 2
  QTcF, Day 113, n=5,6,3,4,2 | -1.08 (20.24) | -1.0 (14.09) | 4.0 (12.29) | -6.5 (10.75) | -7.0 (5.66)

27. Secondary Outcome: Change From Baseline in Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Viral Load in Plasma at Day 29
Description: Blood samples were collected from participants to assess HBV DNA viral load. Baseline is the last non-missing measurement prior to the first dose of study drug. The concentrations were logarithmic transformed with base 10 in this analysis. Change from Baseline is defined as post-dose visit value minus Baseline value. The last observation carried forward (LOCF) method was used to impute missing values at Day 29 in this analysis.
Time Frame: Baseline (Day 1 pre-dose) and Day 29
Population: Full Analysis Set Population comprised of practically-feasible Intent-to-treat population, including subset of the Safety Set with a Baseline and at least 1 post-Baseline plasma HBV DNA concentration. Only those participants with data available at the specified data points were analyzed. In Cohort 3 participants were administered GSK3228836 300 mg instead of 450 mg as per sponsor's decision,hence Cohort 2 and Cohort 3 have been combined.
Measure: Mean (Standard Deviation); unit: Log10 (International Units/milliliter)
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Log10 (International Units/milliliter) | -0.384 (0.4199) | -1.655 (1.4791) | -0.001 (0.4710) | 0.075 (0.1667) | 0.000 (0.0000)
Statistical Analysis 1: Comparison: Cohort 1 GSK3228836 150 mg vs Cohorts 1-3 Placebo; Test type: Other; p = 0.116, ANCOVA — Baseline was the covariate and treatment group as a factor for the comparison between GSK3228836 and placebo group
Statistical Analysis 2: Comparison: Cohort 2 and Cohort 3 GSK3228836 300 mg vs Cohorts 1-3 Placebo; Test type: Other; p < 0.001, ANCOVA — Baseline was the covariate and treatment group as a factor for the comparison between GSK3228836 and placebo group
Statistical Analysis 3: Comparison: Cohort 4 GSK3228836 300 mg vs Cohort 4 Placebo; Test type: Other; p = 0.573, ANCOVA — Baseline was the covariate and treatment group as a factor for the comparison between GSK3228836 and placebo group

28. Secondary Outcome: Change From Baseline in Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Viral Load in Plasma at Week 31
Description: Blood samples were collected from participants to assess HBV DNA viral load. Baseline is the last non-missing measurement prior to the first dose of study drug. The concentrations were logarithmic transformed with base 10 in this analysis. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Week 31
Population: Full Analysis Set Population. Only those participants with data available at the specified data points were analyzed. In Cohort 3 participants were administered GSK3228836 300 mg instead of 450 mg as per sponsor's decision, hence Cohort 2 and Cohort 3 have been combined.
Measure: Mean (Standard Deviation); unit: Log10 (International Units/milliliter)
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 5 | 12 | 5 | 3 | 1
Log10 (International Units/milliliter) | -4.754 (0.8344) | -4.770 (1.2823) | -3.547 (1.2798) | 0.000 (0.0000) | 0.000 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
Statistical Analysis 1: Comparison: Cohort 1 GSK3228836 150 mg vs Cohorts 1-3 Placebo; Test type: Other; p = 0.609, ANCOVA — Baseline was the covariate and treatment group as a factor for the comparison between GSK3228836 and placebo group
Statistical Analysis 2: Comparison: Cohort 2 and Cohort 3 GSK3228836 300 mg vs Cohorts 1-3 Placebo; Test type: Other; p = 0.141, ANCOVA — Baseline was the covariate and treatment group as a factor for the comparison between GSK3228836 and placebo group

29. Secondary Outcome: Change From Baseline in HBV Surface Antigen (HBsAg) Level in Serum at Day 29
Description: Blood samples were collected from participants to assess HBsAg level. Baseline is the last non-missing measurement prior to the first dose of study drug. The concentrations were logarithmic transformed with base 10 in this analysis. Change from Baseline is defined as post-dose visit value minus Baseline value. The LOCF method was used to impute missing values at Day 29 in this analysis.
Time Frame: Baseline (Day 1 pre-dose) and Day 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Log10 (International Units/milliliter)
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Log10 (International Units/milliliter) | -0.504 (0.5656) | -1.556 (1.3787) | 0.000 (0.1116) | -1.986 (1.7986) | -0.008 (0.0390)
Statistical Analysis 1: Comparison: Cohort 1 GSK3228836 150 mg vs Cohorts 1-3 Placebo; Test type: Other — Baseline was the covariate and treatment group as a factor for the comparison between GSK3228836 and placebo group; p = 0.245, ANCOVA
Statistical Analysis 2: Comparison: Cohort 2 and Cohort 3 GSK3228836 300 mg vs Cohorts 1-3 Placebo; Test type: Other; p = 0.001, ANCOVA — Baseline was the covariate and treatment group as a factor for the comparison between GSK3228836 and placebo group
Statistical Analysis 3: Comparison: Cohort 4 GSK3228836 300 mg vs Cohort 4 Placebo; Test type: Other; p = 0.762, ANCOVA — Baseline was the covariate and treatment group as a factor for the comparison between GSK3228836 and placebo group

30. Secondary Outcome: Change From Baseline in HBsAg Level in Serum at Week 31
Description: Blood samples were collected from participants to assess HBsAg level. Baseline is the last non-missing measurement prior to the first dose of study drug. The concentrations were logarithmic transformed with base 10 in this analysis. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Week 31
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Log10 (International Units/milliliter)
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 4 | 2
Log10 (International Units/milliliter) | -0.523 (0.9299) | -0.547 (0.6109) | 0.059 (0.3859) | -1.519 (1.4821) | -0.043 (0.0178)
Statistical Analysis 1: Comparison: Cohort 1 GSK3228836 150 mg vs Cohorts 1-3 Placebo; Test type: Other; p = 0.141, ANCOVA — Baseline was the covariate and treatment group as a factor for the comparison between GSK3228836 and placebo group
Statistical Analysis 2: Comparison: Cohort 2 and Cohort 3 GSK3228836 300 mg vs Cohorts 1-3 Placebo; Test type: Other; p = 0.081, ANCOVA — Baseline was the covariate and treatment group as a factor for the comparison between GSK3228836 and placebo group
Statistical Analysis 3: Comparison: Cohort 4 GSK3228836 300 mg vs Cohort 4 Placebo; Test type: Other; p = 0.616, ANCOVA — Baseline was the covariate and treatment group as a factor for the comparison between GSK3228836 and placebo group

31. Secondary Outcome: Percentage of Participants Who Achieved HBsAg Loss at Day 29 and Week 31
Description: Blood samples were collected to evaluate the percentage of participants with HBsAg loss at Day 29 and Week 31. A 'Loss' of HBsAg means antigen is negative. HBsAg Loss percentage is defined as number of participants with HBsAg loss divided by total number of participants assessed multiplied by 100. Baseline is the last non-missing measurement prior to the first dose of study drug.
Time Frame: At Day 29 and Week 31
Population: Full Analysis Set Population. In Cohort 3 participants were administered GSK3228836 300 mg instead of 450 mg as per sponsor's decision, hence Cohort 2 and Cohort 3 have been combined.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 12 | 6 | 5 | 2
Percentage of Participants
  Day 29 | 0 | 16.7 | 0 | 20.0 | 0
  Week 31 | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Percentage of Participants Who Achieved HBV e Antigen (HBeAg) Loss at Day 29 and Week 31 Who Were HBeAg Positive at Baseline
Description: Blood samples were collected to evaluate the percentage of participants with HBeAg loss at Day 29 and Week 31. A 'Loss' of HBeAg means antigen is negative. HBeAg Loss percentage is defined as number of participants with HBeAg loss divided by number of participants with positive HBeAg at Baseline multiplied by 100. Baseline is the last non-missing measurement prior to the first dose of study drug. Participants was considered HBeAg positive at Baseline if the Baseline value> 0.09 U/mL.
Time Frame: Baseline (Day 1, Pre dose) and at Day 29 and Week 31
Population: Full Analysis Set Population. Only those participants with data available at the specified data points were analyzed. None of the participants were HBeAg positive at Baseline in Cohort 4, hence no data to report (N=0) for Cohort 4 arms. In Cohort 3 participants were administered GSK3228836 300 mg instead of 450 mg as per sponsor's decision, hence Cohort 2 and Cohort 3 have been combined.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 5 | 6 | 2 | 0 | 0
Percentage of Participants
  Day 29 | 0 | 0 | 0 |  |
  Week 31 | 0 | 0 | 0 |  |

33. Secondary Outcome: Change From Baseline in Serum HBeAg Concentration at Day 29 in Participants Who Were HBeAg Positive at Baseline
Description: Blood samples were collected from participants to assess HBeAg level. Baseline is the last non-missing measurement prior to the first dose of study drug. The concentrations were logarithmic transformed with base 10 in this analysis. Change from Baseline is defined as post-dose visit value minus Baseline value. Participant was considered HBeAg positive at Baseline if the Baseline value> 0.09 International Units/milliliter (IU/mL).
Time Frame: Baseline (Day 1, Pre dose) and at Day 29
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Log10 (IU/mL)
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 5 | 6 | 2 | 0 | 0
Log10 (IU/mL) | -0.004 (0.3967) | -0.052 (0.6741) | 0.133 (0.2884) |  |
Statistical Analysis 1: Comparison: Cohort 1 GSK3228836 150 mg vs Cohorts 1-3 Placebo; Test type: Other; p = 0.763, ANCOVA — Baseline was the covariate and treatment group as a factor for the comparison between GSK3228836 and placebo group
Statistical Analysis 2: Comparison: Cohort 2 and Cohort 3 GSK3228836 300 mg vs Cohorts 1-3 Placebo; Test type: Other; p = 0.804, ANCOVA — Baseline was the covariate and treatment group as a factor for the comparison between GSK3228836 and placebo group

34. Secondary Outcome: Change From Baseline in Serum HBeAg Concentration at Week 31 in Participants Who Were HBeAg Positive at Baseline
Description: Blood samples were collected from participants to assess HBeAg level. Baseline is the last non-missing measurement prior to the first dose of study drug. The concentrations were logarithmic transformed with base 10 in this analysis. Change from Baseline is defined as post-dose visit value minus Baseline value. Participant was considered HBeAg positive at Baseline if the Baseline value> 0.09 U/mL.
Time Frame: Baseline (Day 1, Pre dose) and Week 31
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
Number analyzed (Participants) | 5 | 6 | 2 | 0 | 0
Log10 IU/mL | -0.577 (1.3711) | -0.195 (0.5047) | 0.131 (0.7477) |  |
Statistical Analysis 1: Comparison: Cohort 1 GSK3228836 150 mg vs Cohorts 1-3 Placebo; Test type: Other; p = 0.372, ANCOVA — Baseline was the covariate and treatment group as a factor for the comparison between GSK3228836 and placebo group
Statistical Analysis 2: Comparison: Cohort 2 and Cohort 3 GSK3228836 300 mg vs Cohorts 1-3 Placebo; Test type: Other; p = 0.954, ANCOVA — Baseline was the covariate and treatment group as a factor for the comparison between GSK3228836 and placebo group

35. Secondary Outcome: Plasma Concentrations of GSK3228836 in Participants With Chronic HBV Infection
Description: Plasma samples were collected from participants with chronic HBV infection at indicated time points for pharmacokinetic analysis of GSK3228836.
Time Frame: Day 1:pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, and 6 hours post-dose, Days 2 and 23: 24 hours post-dose, Day 4: 72 hours post-dose, Days 8 and 15: pre-dose, Day 22: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, and 6 hours post-dose, and Days 29, 36, 57, 85, 113, and 211
Population: Pharmacokinetic Population consisted of participants who were randomized, received at least 1 dose of study drug, and had at least 1 valid pharmacokinetic metric. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). In Cohort 3 participants were administered GSK3228836 300 mg instead of 450 mg as per sponsor's decision, hence Cohort 2 and Cohort 3 have been combined.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohort 4 GSK3228836 300 mg
Number analyzed (Participants) | 6 | 12 | 5
Nanogram per milliliter
  Day 1, pre-dose, n=6,12,5 | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Day 1, 0.5 hour post-dose, n=6,12,5 | 1187.00 (1052.256) | 2145.58 (1295.533) | 1630.00 (539.583)
  Day 1, 1 hour post-dose, n=6,11,5: number analyzed (Participants) | 6 | 11 | 5
  Day 1, 1 hour post-dose, n=6,11,5 | 1909.33 (1287.383) | 4950.91 (2025.302) | 4074.00 (1314.565)
  Day 1, 1.5 hours post-dose, n=6,12,5 | 2440.00 (1515.823) | 6536.67 (2710.704) | 6100.00 (1816.631)
  Day 1, 2 hours post-dose, n=6,12,5 | 2976.67 (1444.793) | 8387.50 (3287.981) | 7556.00 (2672.579)
  Day 1, 3 hours post-dose, n=6,12,5 | 3360.00 (1614.955) | 9905.00 (3494.308) | 8916.00 (2541.324)
  Day 1, 4 hours post-dose, n=6,12,5 | 3340.00 (1223.781) | 9658.33 (3612.189) | 9632.00 (2115.401)
  Day 1, 5 hours post-dose, n=6,12,5 | 3210.00 (1156.962) | 9813.33 (3524.376) | 9122.00 (2616.662)
  Day 1, 6 hours post-dose, n=6,12,5 | 2933.33 (986.097) | 9345.00 (3258.863) | 8580.00 (2203.418)
  Day 2, 24 hours post dose, n=6,12,5 | 112.22 (79.406) | 336.88 (301.302) | 356.00 (140.490)
  Day 4 , 72 hours post-dose, n=6,12,5 | 6.77 (2.759) | 12.92 (3.975) | 15.24 (3.138)
  Day 8, pre-dose, n=6,12,4: number analyzed (Participants) | 6 | 12 | 4
  Day 8, pre-dose, n=6,12,4 | 7.69 (4.540) | 22.07 (7.715) | 21.80 (6.458)
  Day 15, pre-dose, n=6,12,4: number analyzed (Participants) | 6 | 12 | 4
  Day 15, pre-dose, n=6,12,4 | 10.90 (4.989) | 30.29 (12.598) | 33.33 (11.536)
  Day 22, pre-dose, n=5,12,4: number analyzed (Participants) | 5 | 12 | 4
  Day 22, pre-dose, n=5,12,4 | 9.38 (2.279) | 22.85 (9.848) | 25.43 (7.630)
  Day 22 0.5 hour pre-dose, n=5,12,4: number analyzed (Participants) | 5 | 12 | 4
  Day 22 0.5 hour pre-dose, n=5,12,4 | 1315.40 (1064.380) | 2073.58 (883.806) | 1447.75 (850.592)
  Day 22, 1 hour post-dose, n=5,12,4: number analyzed (Participants) | 5 | 12 | 4
  Day 22, 1 hour post-dose, n=5,12,4 | 2133.00 (1616.738) | 4815.83 (1835.595) | 3477.50 (2009.766)
  Day 22, 1.5 hours post-dose, n=5,12,4: number analyzed (Participants) | 5 | 12 | 4
  Day 22, 1.5 hours post-dose, n=5,12,4 | 2874.00 (1872.173) | 7094.17 (2862.178) | 5235.00 (3036.341)
  Day 22, 2 hours post-dose, n=5,12,4: number analyzed (Participants) | 5 | 12 | 4
  Day 22, 2 hours post-dose, n=5,12,4 | 3466.00 (2033.158) | 8351.67 (3274.596) | 6765.00 (3805.422)
  Day 22, 3 hours post-dose, n=5,12,4: number analyzed (Participants) | 5 | 12 | 4
  Day 22, 3 hours post-dose, n=5,12,4 | 4070.00 (2146.742) | 9137.50 (3303.139) | 8325.00 (5007.950)
  Day 22, 4 hours post-dose, n=5,12,4: number analyzed (Participants) | 5 | 12 | 4
  Day 22, 4 hours post-dose, n=5,12,4 | 3760.00 (1572.260) | 8650.00 (2913.339) | 8690.00 (4808.791)
  Day 22, 5 hours post-dose, n=5,12,4: number analyzed (Participants) | 5 | 12 | 4
  Day 22, 5 hours post-dose, n=5,12,4 | 3566.00 (1229.504) | 8072.50 (2748.322) | 8027.50 (4274.166)
  Day 22, 6 hours post-dose, n=5,12,4: number analyzed (Participants) | 5 | 12 | 4
  Day 22, 6 hours post-dose, n=5,12,4 | 2990.00 (817.099) | 7769.17 (2295.697) | 7447.50 (3817.376)
  Day 23, 24 hours post-dose, n=5,12,4: number analyzed (Participants) | 5 | 12 | 4
  Day 23, 24 hours post-dose, n=5,12,4 | 152.90 (148.879) | 387.88 (209.944) | 524.00 (372.305)
  Day 29, n=5,12,4: number analyzed (Participants) | 5 | 12 | 4
  Day 29, n=5,12,4 | 8.88 (1.680) | 23.42 (9.358) | 21.50 (4.883)
  Day 36, n=5,12,4: number analyzed (Participants) | 5 | 12 | 4
  Day 36, n=5,12,4 | 5.32 (1.098) | 12.58 (6.332) | 8.96 (3.246)
  Day 57, n=5,12,4: number analyzed (Participants) | 5 | 12 | 4
  Day 57, n=5,12,4 | 1.91 (0.405) | 3.80 (1.294) | 1.90 (0.752)
  Day 85, n=5,12,4: number analyzed (Participants) | 5 | 12 | 4
  Day 85, n=5,12,4 | 0.00 (0.00) | 1.32 (0.872) | 0.31 (0.625)
  Day 133, n=5,12,4: number analyzed (Participants) | 5 | 12 | 4
  Day 133, n=5,12,4 | 0.91 (1.273) | 0.59 (0.619) | 0.00 (0.00)
  Day 211, n=5,12,4: number analyzed (Participants) | 5 | 12 | 4
  Day 211, n=5,12,4 | 0.38 (0.845) | 1.04 (2.438) | 0.37 (0.730)

ADVERSE EVENTS:
Time Frame: Non-serious (>=5%) and serious adverse events were collected up to Day 211
Description: Non-serious and serious adverse events were collected in the Safety Population. In Cohort 3 participants were administered GSK3228836 300 mg instead of 450 mg as per sponsor's decision, hence Cohort 2 and Cohort 3 have been combined.
Arm/Group | Cohort 1 GSK3228836 150 mg | Cohort 2 and Cohort 3 GSK3228836 300 mg | Cohorts 1-3 Placebo | Cohort 4 GSK3228836 300 mg | Cohort 4 Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/12 | 0/6 | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/12 | 0/6 | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 5/6 | 6/12 | 2/6 | 3/5 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 GSK3228836 150 mg (N=6) | Cohort 2 and Cohort 3 GSK3228836 300 mg (N=12) | Cohorts 1-3 Placebo (N=6) | Cohort 4 GSK3228836 300 mg (N=5) | Cohort 4 Placebo (N=2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 GSK3228836 150 mg (N=6) | Cohort 2 and Cohort 3 GSK3228836 300 mg (N=12) | Cohorts 1-3 Placebo (N=6) | Cohort 4 GSK3228836 300 mg (N=5) | Cohort 4 Placebo (N=2)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 3 (9) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 2 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (5) | 1 (1) | 1 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial

DOCUMENTS (2):
  • Study Protocol (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT02981602/Prot_002.pdf
  • Statistical Analysis Plan (2019-12-23): https://cdn.clinicaltrials.gov/large-docs/02/NCT02981602/SAP_001.pdf